CLINICAL TRIAL: NCT05663528
Title: ANALYSIS OF CLINICAL AND LABORATORY VARIABLES WITH PREDICTION CAPABILITY FOR INDICATION OF INVASIVE MECHANICAL VENTILATION IN PATIENTS WITH COVID-19
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, JOSE ROBERTO LAPA E SILVA, MD PhD, Universidade Federal do Rio de Janeiro
Other Study IDs: 100685
Record Dates: First submitted 2022-12-21; First posted 2022-12-23 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: COVID-19
Keywords: mechanical ventilation; Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- orotracheal intubation group: Composed of Patients who were intubated after 48 hours of admission to the intensive care unit
  Interventions: Procedure: orotracheal intubation
- non-intubated group: Composed of patients who were not intubated during their stay in the intensive care unit

INTERVENTIONS:
Procedure: orotracheal intubation — Clinical and laboratory data will be collected from patients who are intubated after 48 hours of admission to the intensive care unit
  Other Names: invasive mechanical ventilation
  Groups: orotracheal intubation group

SUMMARY:
This observational and retrospective study will follow the recommendations of the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE). The aim is to verify and analyze the clinical and laboratory variables with prediction capability for indication of invasive ventilatory support in patients with COVID-19. The present study will be carried out in specific care units for patients with suspected or confirmed COVID-19. Individuals with suspected or clinical diagnosis of COVID-19, with a minimum hospital stay of 24 hours and submitted to oxygen therapy or non-invasive ventilation will be selected. Clinical and laboratory variables will be collected from the moment of admission and every 12 hours until the third day of hospitalization. The primary outcome will be rate of endotracheal intubation, while secondary outocomes will be lenght of stay in intensive care unit, and hospital, as well as mortality rate.

DETAILED DESCRIPTION:
Clinical and laboratory data will be collected from medical records from the period of the COVID-19 pandemic (February 2020 to June 2021)

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be individuals with confirmed diagnosis of COVID-19 by RT-PCR (reverse- transcriptase polymerase chain reaction), with minimum length of stay of 24 hours in the ICU and, patients who sign the free and clarified consent.

Exclusion Criteria:

* The exclusion criteria for participation in the study will be as follows: (1) patients under the age of 18; (2) patients with a negative laboratory test for COVID-19; (3) patients in need of emergency intubation; (4) patients who underwent previous endotracheal intubation at the same hospitalization.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with confirmation of covid-19 and with length of stay in the intensive care unit greater than 48 hours will be selected for the intubated and non-intubated groups. For the intubated group, patients who underwent endotracheal intubation after 48 hours of admission to the intensive care unit will be selected. For the non-intubated group, those patients who were not intubated during their stay in the intensive care unit will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Identify clinical and laboratory variables that may be associated with the need of endotracheal intubation in the first 72 hours of admission to the intensive care unit. | 3 days
  Vital signs will be collected through the cardiac monitor and clinical evaluation from the moment of admission until the third day of hospitalization, every twelve hours and full blood count and biochemistry data will be collected from patients at admission until the third day of hospitalization in the intensive care unit

SECONDARY OUTCOMES:
time to endotracheal intubation | 28 days
  It will be collected from the date of intensive care unit admission until the date of endotracheal intubation
length of stay in the ICU | 6 months
  It will be collected from the date of intensive care unit admission until the outcome of discharge from the intensive care unit or death.
length of hospital | 12 months
  It will be collected from the date of intensive care unit admission until the outcome of hospital discharge or death.
mechanical ventilation days | 6 months
  It will be collected from the date of intubation in the intensive care unit until the date of extubation or up to 48 hours off mechanical ventilation in cases of tracheostomized patients and/or until the outcome of death
hospital mortality | 12 months
  Mortality will be collected during the period of hospitalization

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Pedro Ernesto University Hospital, Rio de Janeiro
  - National Institute of Infectology Evandro Chagas, Rio de Janeiro
  - Clementino Fraga Filho University Hospital, Rio de Janeiro

REFERENCES:
- [Derived] Maia G, Martins CM, Marques V, Christovam S, Prado I, Moraes B, Rezoagli E, Foti G, Zambelli V, Cereda M, Berra L, Rocco PRM, Cruz MR, Samary CDS, Guimaraes FS, Silva PL. Derivation and external validation of predictive models for invasive mechanical ventilation in intensive care unit patients with COVID-19. Ann Intensive Care. 2024 Aug 21;14(1):129. doi: 10.1186/s13613-024-01357-4. PMID 39167241